CLINICAL TRIAL: NCT04502719
Title: Comparison of Two Nutritional Screening Tools for the Detection of Malnutrition in Patients with Liver Cirrhosis
Brief Title: Comparison of Nutritional Screening Tools in Liver Cirrhosis Patients
Status: Recruiting | Type: Observational
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Joan Trabal, RDN, PhD, Hospital Clinic of Barcelona
Other Study IDs: NUSCIR-20
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Malnutrition; Cirrhosis, Liver
Keywords: malnutrition; liver cirrhosis; sarcopenia; quality of life
MeSH Terms: conditions — Malnutrition; Liver Cirrhosis; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Screened: Patients with liver cirrhosis screened for malnutrition.
  Interventions: Diagnostic Test: Nutritional screening.

INTERVENTIONS:
Diagnostic Test: Nutritional screening. — Nutritional screening with the RFH-NPT and LDUST questionnaires.

SUMMARY:
This study compares two nutritional screening questionnaires in cirrhotic patients. All patients will be assessed with both questionnaires, besides a complete nutritional assessment.

DETAILED DESCRIPTION:
Disease-related malnutrition is a health problem with high prevalence and associated costs. Poor nutritional status has an unfavorable effect on clinical outcomes in terms of complications, post-transplant survival and mortality in relation to the liver, in addition to a decrease in quality of life. The same complications of liver disease, such as hypoalbuminemia or ascites, make it difficult to assess malnutrition in cirrhotic patients.

The use of screening tools defines the first step in the prevention and treatment of patients at risk of malnutrition or overt malnutrition. The use of screening tools to detect malnutrition upon admission to hospital improves the identification of malnourished patients by 50-80%, early treatment of patients can reduce hospital stay. It has been observed that nutritional interventions, after assessment of nutritional risk, appear to prevent complications and improve quality of life and survival rate in cirrhotic patients.

Due to changes in body composition in cirrhotic patients (i.e. ascites), the most common questionnaires for screening for malnutrition (e.g. MUST, NRS-2002), which use anthropometric measures, have not been validated in cirrhosis and are therefore not considered suitable for malnutrition screening. On the contrary, in recent years two specific nutritional screening tools have been developed for cirrhotic patients, the Royal Free Hospital Nutritional Prioritizing Tool (RFH-NPT) and the Liver Disease Undernutrition Screening Tool (LDUST). Both questionnaires, however, require further validation against clinical outcomes in cirrhotic patients.

This study will use two screening tools for malnutrition risk (RFH-NPT and LDUST), to compare their validity in detecting malnutrition risk in patients with liver cirrhosis. These tools will be validated by performing a nutritional assessment with the new diagnostic criteria of malnutrition promoted by the Global Leadership Initiative on Malnutrition.

Sarcopenia can occur in malnourished cirrhotic patients, so it will be of interest to know what the possible prevalence may be in the sample of patients studied. The use of the screening questionnaire SARC-F will allow an assessment of the prevalence of risk of sarcopenia. Situations such as malnutrition or sarcopenia can have an impact on the patient's health-related quality of life, so this parameter will be assessed using the Chronic Liver Disease Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with liver cirrhosis.

Exclusion Criteria:

* Patients with cognitive impairment or major psychiatric disorder.
* Lack of consent from the patient for inclusion in the study.
* Any patient who is not suitable based on the researcher's own judgement.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort will be selected from admitted patients at the Hepatology ward of the Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2021-02-22 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Malnutrition diagnostic concordance. | 48 hours
  Diagnostic concordance between nutritional screening questionnaires and nutritional assessment using GLIM criteria

SECONDARY OUTCOMES:
Malnutrition prevalence. | 48 hours.
  Prevalence of malnutrition according to the GLIM criteria.
Sarcopenia prevalence. | 48 hours.
  Prevalence of the risk of sarcopenia assessed with the SARC-F (Strength, Assistance, Rise, Climb-Falls) questionnaire. Minimum and maximum values: 0-10. Higher scores mean a worse outcome.
Quality of life score. | 48 hours.
  Quality of life score according to the Chronic Liver Disease Questionnaire (CLDQ). Minimum and maximum values: 5-36. Higher scores mean a better outcome.
Adverse clinical outcomes. | 6 months.
  Number of adverse clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Joan Trabal, RDN, PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferreira LG, Anastacio LR, Lima AS, Touslon Davisson Correia MI. Predictors of mortality in patients on the waiting list for liver transplantation. Nutr Hosp. 2013 May-Jun;28(3):914-9. doi: 10.3305/nh.2013.28.3.6333. PMID 23848119
- [Background] Iwasa M, Iwata K, Hara N, Hattori A, Ishidome M, Sekoguchi-Fujikawa N, Mifuji-Moroka R, Sugimoto R, Fujita N, Kobayashi Y, Takei Y. Nutrition therapy using a multidisciplinary team improves survival rates in patients with liver cirrhosis. Nutrition. 2013 Nov-Dec;29(11-12):1418-21. doi: 10.1016/j.nut.2013.05.016. PMID 24103520
- [Background] Tandon P, Raman M, Mourtzakis M, Merli M. A practical approach to nutritional screening and assessment in cirrhosis. Hepatology. 2017 Mar;65(3):1044-1057. doi: 10.1002/hep.29003. Epub 2017 Feb 6. PMID 28027577
- [Background] Cederholm T, Jensen GL, Correia MITD, Gonzalez MC, Fukushima R, Higashiguchi T, Baptista G, Barazzoni R, Blaauw R, Coats A, Crivelli A, Evans DC, Gramlich L, Fuchs-Tarlovsky V, Keller H, Llido L, Malone A, Mogensen KM, Morley JE, Muscaritoli M, Nyulasi I, Pirlich M, Pisprasert V, de van der Schueren MAE, Siltharm S, Singer P, Tappenden K, Velasco N, Waitzberg D, Yamwong P, Yu J, Van Gossum A, Compher C; GLIM Core Leadership Committee; GLIM Working Group. GLIM criteria for the diagnosis of malnutrition - A consensus report from the global clinical nutrition community. Clin Nutr. 2019 Feb;38(1):1-9. doi: 10.1016/j.clnu.2018.08.002. Epub 2018 Sep 3. PMID 30181091